CLINICAL TRIAL: NCT01525056
Title: Rectal Cancer: Local Staging, Re-staging and Assessment of Lymph Node Metastases Using PET-CT, CT-Perfusion and 3T MRI: A Prospective Feasibility Study
Brief Title: Rectal Cancer: Local Staging, Re-staging and Assessment of Lymph Nodes Using Pet-Ct, CT-Perfusion and 3T MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Barbara Fisher, Doctor, London Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LRCP01
Record Dates: First submitted 2012-01-25; First posted 2012-02-02 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; imaging; PET; MRI
MeSH Terms: conditions — Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imaging with ct, mri and pet scans (Other): ct,mri and pet scans pre and post radiation
  Interventions: Radiation: ct and mri scans; Radiation: ct, mri and pet scan; Radiation: ct, mri and pet scans

INTERVENTIONS:
Radiation: ct and mri scans — ct and mri scan preradiation and postradiation
Radiation: ct, mri and pet scan — ct, mri and pet scans preradiation and postradiation
Radiation: ct, mri and pet scans — single arm with ct, mri and pet scans pre and post radiation

SUMMARY:
The purpose of this study is to evaluate the accuracy of Positron emission tomography, Computed Tomography perfusion and 3 Tesla MRI in the radiological down-staging of rectal cancer following neoadjuvant chemoradiation. The restaging result obtained by these imaging studies will be compared to standard imaging studies and the histopathology of the surgical specimen. We hypothesize that these 3 imaging modalities will detect lymph node metastases pretreatment better than standard pretreatment scans and will better determine the degree of response of the primary rectal tumor to preoperative chemoradiation.

DETAILED DESCRIPTION:
Patient Recruitment:

30 consecutive patients with histologically-proven, non-mucinous rectal cancer will be recruited and stratified into three separate groups as follows:

* T2 tumors (requiring only surgery)
* Early T3 tumors (requiring preoperative standard course radiation therapy)
* Advanced T3 and T4 tumors (requiring preoperative chemoradiation)

Study Protocol:

The pretreatment imaging studies will be performed with a 3T MRI pelvis,PET-CT and CT-Perfusion of the pelvis. The patient will then receive standard treatment consisting of surgery,radiation therapy or a course of neoadjuvant chemoradiation.For patients with T3 and T4 tumors, repeat imaging using all three modalities outlined above will be performed post-treatment.

Histopathology & data analysis

MRI Protocol:

All patients will be examined on a 3-T MRI unit (Siemens Medical, Germany) at St. Joseph's Hospital, London.

The MRI protocol is as follows:

* Buscopan 40 mg IM/IV prior to study
* Axial T2 TSE of the entire pelvis (aortic bifurcation to pubic symphysis)
* Sagittal T2 TSE (240 cm FOV) for detection of the rectal tumor
* Axial oblique T2 TSE (220 cm FOV) perpendicular to the rectal tumor
* 3 mm slice thickness
* Coronal T2 TSE (220 cm FOV)
* Axial DWI (B values 0, 500, 1000)
* ADC map

Unless otherwise specified, slice thickness is 4mm. Technique is free-breathing; no bowel preparation, intraluminal or intravascular contrast agents are administered.

PET-CT Protocol:

* Patient fasts for 6-12 hours prior to study, depending on timing of scan
* Patients to be scanned in the morning will fast overnight; those being scanned in the afternoon will fast for 6 hours following a light breakfast.
* Blood sugar level measurement prior to study (should be less than 11 mmol/L). Insulin dependent diabetics are scanned in the early afternoon following a light breakfast and routine morning insulin.
* Exclude pregnancy with urine/serum hCG
* Intravenous injection of 5MBq/kg of F-18 FDG)
* Intravenous injection of 20 mg Lasix, 10 minutes following F-18 FDG injection
* IV hydration with 250-500 mL of saline
* 60 minutes post-injection, acquire non contrast CT and positron emission tomography imaging of the pelvis

CT Perfusion Protocol:

All patients will undergo CT Perfusion with a 64-slice CT scanner (Discovery CT750 HD, GE Healthcare) at St. Joseph's Health Care, London.

The protocol is as follows:

* Preliminary non-contrast 2.5-mm-thick helical CT of the pelvic region (from the aortic bifurcation to the symphysis pubis) with free-breathing to locate a 8-cm section of the rectal tumor that was imaged in the MRI study.
* Prescribe a CT Perfusion study using the axial shuttle mode on the 8-cm section identified above. The perfusion study consists of two phases. The selected pelvic section is scanned every 2.8 s for 64.4 s (24 times) in the first phase and every 15 s for the next 120 s (8 times) in the second phase. The total duration of scanning is 184.4 s. The scanning parameters for both phases are: 120 kVp, 125 mA, 0.4 s rotation period, and 5 mm thick slices. All dynamic images will be reconstructed with adaptive statistical iterative reconstruction (ASIR) technique to reduce noise.
* Contrast injected at a rate of 3-4 ml/s will start at the same as the two-phase scanning, to allow for acquisition of 3-4 baseline volumes (before contrast arrives in the pelvis).
* Free-breathing is allowed during scanning.
* Contrast dose is 0.8ml/kg of body weight up to maximum of 70 ml of contrast at a concentration of 370 mg iodine/ml.
* The acquired dynamic contrast enhanced (DCE) images will be analyzed by CT Perfusion (GE Healthcare) to determine blood flow, blood volume, mean transit time and capillary permeability surface area of the tumor.

Surgical Resection and histopathological examination:

* Total mesorectal excision as per standardized surgical technique; orientation of surgical specimen according to pre-established regional lymph node map -Mapping of regional lymph nodes by pathologist into perirectal zones (anterior, posterior, left, right, superior, middle, inferior)
* Compare pre- and post-therapeutic imaging with histopathological findings.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer, stage T2, T3, T4

Exclusion Criteria:

* Rectal cancer, stage T1 or metastatic
* Non-rectal primary cancer invading the rectum
* Mucinous histology
* Patient is initially, or becomes a non-surgical candidate during the course of the study
* Hip prosthesis (affects PET-CT image processing)
* Allergy to CT contrast or patients with impaired renal function, defined as estimated glomerular filtrate rate (eGFR)< 30 ml/min
* Prior radiotherapy to the region of the study that would result in overlap of radiation fields
* Contraindications to MRI
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
efficacy of PET, CT-perfusion and MRI to stage patients with rectal cancer | 3 years
  The patient will undergo imaging studies with PET, CT-perfusion and MRI before and after standard preoperative chemoradiation and these imaging studies will be compared with standard imaging and with the final pathology specimen in order to determine the accuracy of these 3 studies in detecting lymph node metastases and response of the primary tumour to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Fisher, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada